CLINICAL TRIAL: NCT05477927
Title: A Phase Ia/Ib, Open-label, Single-arm, Dose-escalation and Expansion Study of Specific Dual-targeting VEGFR1 and PD-L1 CAR-T in Cancer Patients With Pleural or Peritoneal Metastases
Brief Title: Dual-targeting VEGFR1 and PD-L1 CAR-T for Cancers Patients With Pleural or Peritoneal Metastases
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Director of Institute of Drug Clinical Trial of West China Hospital, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCART-006
Record Dates: First submitted 2022-05-07; First posted 2022-07-28 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Malignant Peritoneal Effusion; Malignant Ascites; Serous Cavity Metastatises
Keywords: CAR-T regional injection; Solid Tumors; Serosal Cavity metastases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T cell therapy (Experimental): Dual-targeting VEGFR1 and PD-L1 CAR-T cells
  Interventions: Biological: Dual-targeting VEGFR1 and PD-L1 CAR-T cells

INTERVENTIONS:
Biological: Dual-targeting VEGFR1 and PD-L1 CAR-T cells — In the dose escalation part, the dose levels will be escalated following a traditional escalation scheme for 3+3 design.
  In the dose expansion part, patients will be assigned to different groups based on pleural or peritoneal metastases condition.

SUMMARY:
Serosal cavity metastases of malignant tumor seriously affects the quality of life and survival time of patients with cancers in advanced stage. VEGFR1 is frequently expressed in breast cancer, ovarian cancer, lung cancer, gastric cancer and other malignant tumors and their metastases. The VEGFR1/PD-L1 dual-targeting CAR-T will be investigated in cancer patients with serosal cavity metastases.

DETAILED DESCRIPTION:
In this study, VEGFR1 will be used as the general target of serosal cavity metastasis of malignant tumor, and the dual-targeting CAR-T of VEGFR1/PD-L1 will be injected in to pleural or peritoneal cavity of patients with advanced serous cavity metastases, such as ovarian cancer, breast cancer, lung cancer and gastric cancer, who had nearly no response to standard treatment. The safety and effectiveness will be evaluated. The safety evaluation standard refers to the standard of CTCAE 5.0. The evaluation standard of effectiveness refers to the evaluation standard of solid tumor curative effect RECIST 1.1 to evaluate the curative effect.

There are two part of this study, the first is dose escalation part, 18 patients with malignant tumor (failure of standard treatment will be enrolled at least, patients with peritonea cavity metastases are planned to be enrolled in the cohort 1, and those with pleural cavity metastasis are enrolled in the cohort 2. The second is dose expansion part, the curative effect has observed in the first part, and after the DLT observation period of the related dose group was finished, the PI will decided whether to conduct the dose expansion research finally. It was planned to enroll 40 patients with serous cavity metastases , two cohorts were divided the same as mentioned above in dose escalation part.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age 18-65 years old; negative results of serum or urine pregnancy test within 48 hours before treatment are needed to provide for fertile women (or women who have undergone sterilization or at least 2 years after menopause can be regarded as infertile);
2. Patients diagnosed as ovarian cancer, non-small cell lung cancer, breast cancer, gastric cancer, etc., accompanied by serous cavity metastasis, have received systemic standard treatment, and have clinical symptoms of serous cavity metastasis;
3. The Eastern Cooperative Oncology Group (ECOG) performance status score is 0-2;
4. Estimated life expectancy ≥ 3 months (according to investigator's judgement);
5. Absolute neutrophil count ≥ 1.5×10^9/L, platelet count ≥ 90×10^9/L, absolute lymphocyte count ≥1×10^8/L, hemoglobin ≥ 9.0 g/dL;
6. Creatinine clearance rate ≥60 mL/min, Serum ALT/AST≤2.5 times of the normal level, and total bilirubin≤1.5 times of the normal level;
7. Cardiac ejection fraction ≥50%, no pericardial effusion;
8. No other serious diseases (autoimmune diseases or any immune deficiency disease or other disease in need of immunosuppressive therapy);
9. Patients must stop chemotherapy and targeted therapy for at least 3 weeks before starting treatment;
10. Patients must take reliable contraceptive measures before entering the trial, during the research process until 1 year after CAR-T infusion; reliable contraceptive measures will be determined by the main investigator or designated personnel;
11. Voluntarily participate in the research, understand and sign the informed consent;
12. The side effect of the last anti-tumor treatment was reduced to ≤1 grade, except for hair loss.

Exclusion Criteria:

1. Had accepted any treatment of CAR-T therapy;
2. Allergic to cytokines; uncontrolled activity infection;
3. Acute or chronic (graft-versus-host disease) GVHD;
4. Accompanied by other uncontrolled malignant tumors;
5. Patient with hepatitis B or C active period, HIV infection ≥ the upper limit of the normal level;
6. Other uncontrolled diseases in active period that hinder participation in the trial;
7. Suffer from serious diseases such as coronary heart disease, angina pectoris, myocardial infarction, arrhythmia, cerebral thrombosis, cerebral hemorrhage, etc.;
8. Patients with grade 2-3 hypertension or poorly controlled;
9. History of mental illness that is difficult to control;
10. Patients have used immunosuppressive agents for a long time after organ transplantation, except for recent or current inhaled corticosteroid therapy;
11. The existing medical history or mental state history or laboratory abnormalities may increase the risk associated with participating in the study or the administration of the study drug from the point view of PI;
12. Unstable pulmonary embolism, deep venous embolism or other major arterial/venous thromboembolic events occurred within 6 months before enrollment. If receiving anticoagulant therapy;
13. Pregnant or nursing women, or plan to become pregnant during the treatment period or within 1 year after the treatment ends;
14. Female subjects of childbearing age were reluctant to accept high-efficiency contraceptive measures during the treatment period or within 1 year after the treatment ends;
15. Patient suffering from diseases that have signed written informed consent or comply with research procedures; or are unwilling or unable to comply with research requirements;
16. Patients who are inappropriate to participate in this experiment as considered by PI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2023-11-28 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
AEs will be recorded and evaluated by CTCAT 5.0. | 28 days
  Safety
Recommended phase II dose (RP2D). | Approximately 18 months.
  Efficacy dose
Therapeutic efficacy will be evaluated according to RECIST1.1. | Approximately 18 months.
  Ant-tumor effects
Dose-limiting toxicity (DLT) will be assessed by CTCAE 5.0. | 28 days
  Tolerability evaluation

SECONDARY OUTCOMES:
Objective Remission Rate (ORR). | 3 months
  Include CR (complete response) and PR (partial response).
Progression-Free Survival (PFS ). | Approximately 18 months.
  The time from CAR-T administration to disease progression or death.
Duration Of Control Rate (DCR). | 3 months
  The number of cases in which response (PR + CR) and stable disease (SD) are achieved from the start of cell infusion/the total number of evaluable cases (%).
Duration Of Response (DOR). | Approximately 18 months.
  It refers to the time from the first evaluation of CR or PR to the first evaluation of PD(Progressive Disease) or death from any reason.
Overall-Survival (OS). | Approximately 18 months.
  It defined as the time from randomization to death from any cause, is a direct measure of clinical benefit to a patient. Patients alive or lost to follow-up are censored.
Anti-CAR antibody production | 12 months.
  Immunogenicity
CAR-T cell numbers. | 12 months.
  PK/PD

CONTACTS AND LOCATIONS:
Overall Officials: YongShen Wang, Prof., Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

REFERENCES:
- [Background] Cheema PK, Burkes RL. Overall survival should be the primary endpoint in clinical trials for advanced non-small-cell lung cancer. Curr Oncol. 2013 Apr;20(2):e150-60. doi: 10.3747/co.20.1226. PMID 23559882
- [Background] Wagner DL, Fritsche E, Pulsipher MA, Ahmed N, Hamieh M, Hegde M, Ruella M, Savoldo B, Shah NN, Turtle CJ, Wayne AS, Abou-El-Enein M. Immunogenicity of CAR T cells in cancer therapy. Nat Rev Clin Oncol. 2021 Jun;18(6):379-393. doi: 10.1038/s41571-021-00476-2. Epub 2021 Feb 25. PMID 33633361